CLINICAL TRIAL: NCT03525938
Title: Transversus Abdominis Plane Block for Chronic Postsurgical Orchalgia: SHAM Controlled, Randomized Trial, Three Months Results
Brief Title: Transversus Abdominis Plane Block for Chronic Postsurgical Orchalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Diab Fuad Hetta, Assuit university, south egypt cancer institute, anesthesia department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SECI-IRB-IORG0006563-533
Record Dates: First submitted 2018-04-29; First posted 2018-05-16 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Chronic Post-surgical Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP group (Active Comparator)
  Interventions: Procedure: TAP block
- SHAM group (Sham Comparator)
  Interventions: Procedure: TAP block

INTERVENTIONS:
Procedure: TAP block — Whilst the patient is in the supine position, a high frequency ultrasound probe (10 MH) is placed transverse to the abdominal wall between the costal margin and iliac crest. The needle is introduced in plane of the ultrasound probe directly under the probe and advanced until it reaches the plane between the internal oblique and transversus abdominis muscles. Upon reaching the plane, 2 ml of saline is injected to confirm correct needle position after which 20 ml of levobupivacaine, 25% plus triamcinolone, 80 mg solution is injected for TAP group and 20 ml of saline only is injected for SHAM group.. The transversus abdominis plane is visualized expanding with the injection ( appears as a hypoechoic space)

SUMMARY:
the study will evaluate the effect of transversus abdominis plane block (TAP) on chronic post-groin surgeries orchalgia (chronic testicular pain)

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were patients with chronic scrotal pain (orchialgia) that fulfilled the following criteria:

  1. pain intensity ≥ 5 on the visual analog scale (VAS),
  2. pain that lasted for more than 3 months after groin surgeries,
  3. failed conservative treatment with nonsteroidal anti-inflammatory drugs (NSAIDs)

Exclusion Criteria:

* The exclusion criteria were:

  1. patients with other causes of scrotal pain, e.g., epididymitis, orchitis, and hydrocele,
  2. patients complaining of groin infection and coagulopathy,
  3. patients suffering from hypertension, ischemic heart disease, or psychiatric disorders

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-10-15 (Estimated); Study Completion 2019-11-25 (Estimated)

PRIMARY OUTCOMES:
The change of intensity of pain measured by Visual Analogue Pain (VAS ) score | The pain assessment will be done one month, 2 month and 3 month postprocedure.
  The Visual Analogue Pain (VAS) scale is a tool for intensity of pain scored from 0 to 10, where 0 = no pain and 10 = the worst pain imaginable

CONTACTS AND LOCATIONS:
Locations (1):
- Diab, Asyut, Assuit, Egypt